CLINICAL TRIAL: NCT05618353
Title: Impact of Colchicine on Peri-Operative Major Adverse Cardiovascular Events in Patients With Prior Coronary Revascularization
Brief Title: The Peri-OPerative COlchicine to Reduce Negative Events (POPCORN) Trial
Acronym: POPCORN
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: NYU School of Medicine (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CARA-003-22S; I01CX002358-01A2 (NIH)
Record Dates: First submitted 2022-11-03; First posted 2022-11-16 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; Non-cardiac surgery; Colchicine; Inflammation; Major adverse cardiovascular events
MeSH Terms: conditions — Coronary Artery Disease; Inflammation | interventions — Colchicine

STUDY DESIGN:
Intervention Model Description: One day before surgery: Colchicine 1.2 mg with 0.6 mg PO one hour later. This load will be followed by colchicine 0.6 mg twice daily for a total of 14 days. If a patient is unable to take oral medications (by mouth or nasogastric tube) post-operatively (e.g., post abdominal surgery), colchicine will be held until the clinically treating physician allows resumption of oral medications if still within 14 days post-operation.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Matching placebo at the same time points as the intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Colchicine (Active Comparator): One day before surgery: Colchicine 1.2 mg with 0.6 mg PO one hour later. This load will be followed by colchicine 0.6 mg twice daily for a total of 14 days.
  Interventions: Drug: Colchicine
- Placebo (Placebo Comparator): Matching placebo at same time points as active comparator
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Colchicine — 0.6 mg tablets
  Other Names: Colcrys
  Arms: Colchicine
Drug: Placebo — Matching placebo
  Arms: Placebo

SUMMARY:
Heart disease remains the leading cause of death in Veterans. Inflammation in the arteries of the heart may increase the risk of cardiac death. Patients with heart disease undergoing major surgery are at increased risk of complications after surgery, including heart attack, stroke, and death. The proposed research seeks to better understand the role of inflammation in the damage to the heart and blood vessels after major surgery. This research also seeks to identify the potential beneficial role of a safe medication, colchicine, which has direct effects on inflammatory cells and has been used in the treatment of inflammatory diseases for more than 2000 years, on reducing the rate of complications after surgery. With its quick onset of action and excellent safety profile, colchicine may have the potential to reduce risk of heart injury, stroke, or death after major surgery.

DETAILED DESCRIPTION:
Patients with prior coronary revascularization have a high risk of major adverse cardiovascular events (MACE) after major surgery, up to more than 2-fold when compared to patients without prior coronary revascularization. The pro-inflammatory and hypercoagulable states induced by surgery and the hemodynamic changes caused by fluid shifts and anesthesia are all important triggers of perioperative myocardial ischemia. Indeed, peri-operative systemic inflammation is associated with a nearly 4-fold increase in the risk of perioperative MACE. Neutrophils, the most abundant of inflammatory cells, adhere to inflamed or injured endothelium, migrate into the vessel wall, release proteolytic enzymes that can lead to erosion or rupture of plaque. Peri-operative cytokine generation may also activate the inflammasome and, thereby, macrophage-mediated synthesis of interleukin (IL)-1 , a known target for therapy for secondary prevention of MACE, particularly in the setting of high C-reactive protein (CRP) concentration.

Colchicine is a safe, well-tolerated anti-inflammatory agent that preferentially accumulates in neutrophils compared with other inflammatory cells. Colchicine inhibits chemotaxis, endothelial adhesion, and extravasation of neutrophils at sites of endothelial injury or inflammation; suppresses the inflammasome-mediated production of IL-1 by macrophages; and reduces inflammation and MACE in patients with cardiovascular disease. The Colchicine Cardiovascular Outcomes Trial and Low Dose Colchicine 2 Trial demonstrated a reduction in MACE with colchicine in about 4000 patients with prior myocardial infarction and about 5000 patients with stable coronary artery disease, respectively. The Colchicine-PCI trial demonstrated for the first time that administration of colchicine prior to injury dampens the inflammatory response measured by CRP. The effects of colchicine on peri-operative MACE in patients with prior coronary revascularization or high coronary atherosclerotic burden undergoing major surgery, remains unknown.

The aims of this trial are to 1) assess the effect of colchicine compared to placebo on peri-operative MACE in response to intermediate- or high-risk non-cardiac surgery in patients with prior coronary revascularization or high coronary atherosclerotic burden; 2) characterize the level of systemic inflammation and profile of peri-operative neutrophils in this population; and 3) determine the clinical and genetic predictors of peri-operative MACE and examine factors that determine heterogeneity of treatment response in this population. This prospective, double-blinded, placebo-controlled, randomized trial will enroll 700 participants with prior coronary revascularization or high coronary atherosclerotic burden who undergo intermediate- or high-risk non-cardiac surgery across six VA medical centers that serve as cardiovascular referral centers for their VISNs. Following referral for surgery, and confirmation that the patient meets all study entry criteria, participants will be consented and randomized 1:1 within center to a loading dose of colchicine or placebo one day before surgery and twice daily dosing for 14 days post-operation. DNA will be collected at baseline, while measures of systemic inflammation will be collected at baseline, one day, two days, and at 14 days post-operation (or hospital discharge, whichever occurs earlier). Follow-up for all randomized participants who undergo surgery will occur at 30 days + 7 days.

ELIGIBILITY:
Inclusion Criteria:

Men and women with

* Prior coronary revascularization (via PCI or coronary artery bypass graft surgery) or high coronary atherosclerotic burden (>70% let main disease or >80% disease in the proximal or mid LAD, prox Cx, or prox or mid RCA on coronary angiography), AND
* Referred for intermediate- or high-risk surgery (general abdominal or intraperitoneal surgery, neurosurgery, suprainguinal surgery, peripheral vascular surgery, thoracic surgery).
* If planned for only a laparoscopic or endovascular approach (this includes a minimally invasive hybrid approach such as transcarotid artery revascularization), at least one component of the Revised Cardiac Risk Index score (history of myocardial infarction, history of congestive heart failure, history of transient ischemic attack or stroke, pre-operative use of insulin, pre-operative creatinine >2 mg/dL) should be present.

Exclusion Criteria:

* Colchicine use within one month or history of colchicine intolerance
* Inflammatory bowel disease with history of diarrhea as presentation or chronic diarrhea
* Pre-existent progressive neuromuscular disease

  * amyotrophic lateral sclerosis
  * hereditary muscular disorders
  * myositis
  * necrotizing myopathy
  * myasthenia gravis
  * lambert-eaton syndrome
* Glomerular filtration rate <30mL/minute or on dialysis
* History of cirrhosis, chronic active hepatitis or severe hepatic disease
* History of myelodysplasia with current evidence of cytopenia
* Active infection defined as fever >100.4oF or antibiotic use with white blood cell count greater than the upper limit of normal or lower than the lower limit of normal within 24 hours of randomization (major confounder with increased inflammatory markers)
* Undergoing immunosuppressive or immunostimulatory chemo or biologic therapy
* Pregnant (as confirmed by urine or serum test), nursing, or planning to become pregnant during study participation
* Participating in a competing study or unable to consent
* Any significant condition or situation that may put the participant at higher risk, confound the study results, or interfere with adherence to study procedures
* Patients on strong CYP3A4 and/or P-glycoprotein inhibitors (e.g., ritonavir, clarithromycin, diltiazem, verapamil) at baseline will also be excluded due to potential drug interactions

  * However, if one of these medications are started during the post-operative study period, dose adjustments will be made per drug package insert
  * Participants will also be instructed not to drink grapefruit juice while on study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2023-08-21 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular events | 30 days post-operation
  Defined as a composite rate of myocardial injury, non-fatal MI, non-fatal stroke, and all-cause mortality.

SECONDARY OUTCOMES:
rate of myocardial injury | 30 days post-operation
  rate of myocardial injury
rate of non-fatal MI | 30 days post-operation
  rate of non-fatal MI
rate of non-fatal stroke | 30 days post-operation
  rate of non-fatal stroke
rate of all-cause mortality | 30 days post-operation
  rate of all-cause mortality
Unplanned coronary revascularization | 30 days post-operation
  Unplanned coronary revascularization
Prognostic threshold of myocardial injury | 30 days post-operation
  troponin >30 ng/L (high-sensitivity troponin >65 ng/L or absolute change >14 ng/L or 20-65 ng/L with an absolute change of >5 ng/L)
Change in hsCRP | through 14 days post-operation or at hospital discharge, whichever occurs earlier
  between 1) baseline and one day post-operation, and 2) over time including at two days and 14 days post-operation (or hospital discharge, whichever occurs earlier)

CONTACTS AND LOCATIONS:
Overall Officials: Binita Shah, MD, Principal Investigator — VA NY Harbor Healthcare System, New York, NY
Locations (6):
- United States (6):
  - Birmingham VA Medical Center, Birmingham, AL, Birmingham, Alabama
  - VA Long Beach Healthcare System, Long Beach, CA, Long Beach, California
  - VA NY Harbor Healthcare System, New York, NY, New York, New York
  - Durham VA Medical Center, Durham, NC, Durham, North Carolina
  - Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio
  - VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No